CLINICAL TRIAL: NCT01196234
Title: Paclitaxel/Carboplatin (PC) Followed by Gefitinib or Paclitaxel/Carboplatin (PC) in Advanced Non-small Cell Lung Cancer (NSCLC): Randomized Phase II Study
Brief Title: Paclitaxel/Carboplatin (PC) Followed by Gefitinib Versus PC in Advanced Non-small Cell Lung Cancer
Acronym: PRIDE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Sang-We Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC 2009-0677
Record Dates: First submitted 2010-08-09; First posted 2010-09-08 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel/Carboplatin/Gefitinib (Experimental): Paclitaxel/Carboplatin/Gefitinib
  Interventions: Drug: Paclitaxel/Carboplatin/Gefitinib
- Paclitaxel/Carboplatin (Active Comparator): Paclitaxel/Carboplatin
  Interventions: Drug: Paclitaxel/Carboplatin

INTERVENTIONS:
Drug: Paclitaxel/Carboplatin/Gefitinib — paclitaxel (175mg/m2 on day 1)/carboplatin (AUC 5 on day 1)/daily gefitinib 250mg/day during day 2-15
  Arms: Paclitaxel/Carboplatin/Gefitinib
Drug: Paclitaxel/Carboplatin — paclitaxel (175mg/m2 on day 1)/carboplatin (AUC 5 on day 1)
  Arms: Paclitaxel/Carboplatin

SUMMARY:
This study compares paclitaxel/carboplatin (PC) to PC chemotherapy followed by gefitinib for 2 weeks in patients with Non-small Cell Lung Cancer (NSCLC) without epidermal growth factor receptor (EGFR) mutations.

Expanded acronym : [P]aclitaxel/Ca[r]boplatin (PC) followed by Gef[i]tinib in A[d]vanc[e]d Non-small Cell Lung Cancer (NSCLC): Randomized phase II study.

DETAILED DESCRIPTION:
A randomized phase II trial that compares paclitaxel/carboplatin (PC) to PC chemotherapy followed by gefitinib for 2 weeks in patients with NSCLC without EGFR mutations. While previous studies with cytotoxic agents and gefitinib failed to show any benefit, we altered the schedule of administration in hopes to gain synergy between agents.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years of age
* Histologically documented non-small cell lung cancer with metastasis (Stage IV) or locally advanced (Stage IIIB) with malignant effusion.
* At least 1 measurable lesion as defined by RECIST1.0. All target lesions must have a unidirectional diameter of at least 1cm. Baseline measurements must be compared within 4 weeks prior to enrollment.
* ECOG PS 0-2
* At least 1 week since the last radiotherapy. Patients must have recovered from all acute toxicities from radiotherapy.
* Patients must have adequate hematologic, renal and liver function as defined by Hb > 9g/dL, neutrophils > 1000/mm3, platelets > 50,000/mm3, creatinine < 2mg/dL, and AST (SGOT) and/or ALT (SGPT) < 5 x UNL (upper normal limit).
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.
* Written and voluntary informed consent understood, signed and dated.

Exclusion Criteria:

* Patients with tumor harboring EGFR mutation.
* Prior systemic therapy for NSCLC
* Non-smoking patients with adenocarcinoma. But if those patients show wild type EGFR, they are eligible to this study.
* Symptomatic brain metastasis. Brain metastases stable < 2 weeks before dosing or requiring concurrent steroid treatment or with clinical symptoms.
* Major surgery within 3 weeks prior to study enrollment.
* Previous (less than 3 years ago) or current malignancies at sites other than curatively treated in situ carcinoma of cervix, or basal or squamous cell carcinoma of the skin.
* Severe medical illness or active infection that would impair the ability to receive gefitinib.
* Pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-12; Primary Completion 2012-02 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Response Rate | average 6 months

SECONDARY OUTCOMES:
progression free survival | average 2 years
overall survival | average 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sang-We Kim, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Choi YJ, Lee DH, Choi CM, Lee JS, Lee SJ, Ahn JH, Kim SW. Randomized phase II study of paclitaxel/carboplatin intercalated with gefitinib compared to paclitaxel/carboplatin alone for chemotherapy-naive non-small cell lung cancer in a clinically selected population excluding patients with non-smoking adenocarcinoma or mutated EGFR. BMC Cancer. 2015 Oct 22;15:763. doi: 10.1186/s12885-015-1714-y. PMID 26493267